CLINICAL TRIAL: NCT01952119
Title: Effect of a Secure Message Reminder on Hypertension Follow-up at an Integrated Health Care Delivery System
Brief Title: Effect of a Secure Message Reminder on Hypertension Follow-up at an Integrated Health Care System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GA-11AKuo-01
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Hypertension
Keywords: hypertension
MeSH Terms: conditions — Hypertension

ARMS (2):
- Routine Care (No Intervention): Routine care, no intervention
- Secure message reminder (Active Comparator): Will receive a secure message reminder asking subjects to schedule an appointment with their provider or make a nurse visit to follow-up on their blood pressure
  Interventions: Other: Secure message reminder

INTERVENTIONS:
Other: Secure message reminder — Single secure message reminder asking subjects to schedule an appointment with their provider or make a nurse visit to follow-up on their blood pressure
  Arms: Secure message reminder

SUMMARY:
This study will assess whether adding a secure message reminder to routine care improves the percentage of patients who complete a follow-up appointment with a new, documented blood pressure reading.

DETAILED DESCRIPTION:
Hypertension is one of the leading risk factors for cardiovascular disease. Optimizing blood pressure management can help prevent adverse cardiovascular outcomes. The National Committee for Quality Assurance (NCQA) defines blood pressure control as less than 140/90 mmHg. Per this definition, less than half of Americans with hypertension are considered controlled. Literature has been published describing several ways of improving blood pressure management, but results have been variable.

ELIGIBILITY:
Inclusion Criteria:

* Member of Kaiser Permanente Georgia Pharmacy Cardiac Risk Service (PCRS)
* 18-75 years of age
* Enrolled in http://kp.org
* Most recent documented blood pressure is greater than or equal to 140/90 mmHg

Exclusion Criteria:

* Most recent documented blood pressure is greater than or equal to 180/110 mmHg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Appointment with new blood pressure reading | 6 weeks
  Percentage of patients who complete an appointment with a new documented blood pressure reading within six weeks after distributing the secure message reminder

SECONDARY OUTCOMES:
New appointment with new blood pressure reading | 6 weeks
Existing appointment kept with new blood pressure reading | 6 weeks
Change in antihypertensive regimen | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alina Kuo, PharmD, Principal Investigator — Kaiser Permanente Georgia
Locations (1):
- Kaiser Permanente Georgia, Atlanta, Georgia, United States

REFERENCES:
- [Background] Glynn LG, Murphy AW, Smith SM, Schroeder K, Fahey T. Interventions used to improve control of blood pressure in patients with hypertension. Cochrane Database Syst Rev. 2010 Mar 17;(3):CD005182. doi: 10.1002/14651858.CD005182.pub4. PMID 20238338